CLINICAL TRIAL: NCT01177137
Title: Tinnitus Retraining Therapy Trial
Acronym: TRTT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of Alabama, Tuscaloosa (Other); David Grant U.S. Air Force Medical Center (U.S. Federal Agency); 59th Medical Wing (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency); United States Naval Medical Center, Portsmouth (U.S. Federal Agency); Naval Hospital Camp Pendleton (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U01DC007422 (NIH); U01DC007422 (NIH)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Subjective Tinnitus
Keywords: tinnitus; tinnitus retraining therapy; standard of care; directive counseling; sound therapy; tinnitus questionnaire; tinnitus handicap inventory
MeSH Terms: conditions — Tinnitus | interventions — Standard of Care; Directive Counseling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TRT (Experimental): TRT includes treatment with a conventional sound generator (SG) and directive counseling (DC)
  Interventions: Device: Conventional sound generator (SG); Behavioral: Directive Counseling (DC)
- Partial TRT (Other): Partial TRT includes treatment with a placebo sound generator (placebo SG) and directive counseling (DC).
  Interventions: Device: Placebo sound generator (placebo SG); Behavioral: Directive Counseling (DC)
- Standard of Care (SC) (Other): The standard of care arm includes care as typically delivered in US military medical centers
  Interventions: Behavioral: Standard of Care (SC)

INTERVENTIONS:
Device: Conventional sound generator (SG) — Conventional SGs: Tranquil model sound generators (General Hearing Instruments, Inc.) are either inside or outside-the-ear devices that generate low-level noise, which is set at or just below the patient's mixing point (i.e., the noise level that just blends with the study participant's tinnitus)
  Arms: TRT
Device: Placebo sound generator (placebo SG) — Tranquil model placebo sound generators (General Hearing Instruments, Inc.) are either inside or outside-the-ear devices that generate a sound different from the active devices.
  Arms: Partial TRT
Behavioral: Standard of Care (SC) — The standard of care treatment will be similar to that typically provided to patients with severe tinnitus at participating military medical centers and as described in the American Speech-Language-Hearing Association (ASHA) Preferred Practice Patterns in Audiology (ASHA, 2006). Tinnitus management will be based on the patient's complaints, history, audiologic evaluation, and self-assessment. The goal of the tinnitus management is to reduce negative cognitive, affective, physical, and behavioral reactions to tinnitus and to improve the patient's well-being and quality of life. Specific treatment recommendations will be individualized to reflect the participant's concerns and abilities, as well as his or her engagement in the decision-making process regarding treatment options.
  Arms: Standard of Care (SC)
Behavioral: Directive Counseling (DC) — Directive Counseling (DC): two-hour educational session during which the patient is given information regarding the nature of the tinnitus problem and related problems such as hearing loss and sound intolerance; visual aids to review the audiological/tinnitus/ hyperacusis evaluation, provide instruction on anatomy and physiology of hearing and tinnitus, introduce the Jastreboff neurophysiological model of tinnitus and related concepts of habituation, and describe and recommend the use of ST and environmental sound in the habituation process.
  Arms: TRT
Behavioral: Directive Counseling (DC) — Directive Counseling (DC): two-hour educational session during which the patient is given information regarding the nature of the tinnitus problem and related problems such as hearing loss and sound intolerance; visual aids to review the audiological/tinnitus/ hyperacusis evaluation, provide instruction on anatomy and physiology of hearing and tinnitus, introduce the Jastreboff neurophysiological model of tinnitus and related concepts of habituation, and describe and recommend the use of ST and environmental sound in the habituation process.
  Arms: Partial TRT

SUMMARY:
The primary purpose of the Tinnitus Retraining Therapy Trial (TRTT) is to assess the efficacy of tinnitus retraining therapy (TRT) as a treatment for severe debilitating tinnitus. TRT is a non-medical intervention that uses directive counseling (DC) and sound therapy (ST)to habituate the patient's associated negative emotional reactions to tinnitus, its perception, and ultimately, its impact on the patient's life.

DETAILED DESCRIPTION:
The Tinnitus Retraining Therapy Trial (TRTT), funded by the National Institute of Deafness and Other Communication Disorders, is a multi-center randomized clinical trial testing the efficacy of tinnitus retraining therapy (TRT) versus standard-of-care (SC) treatment in individuals who have self-perceived intolerable tinnitus. TRT is a non-medical intervention that uses directive counseling (DC) and low-level sound therapy (ST) achieved through sound generators (SGs) to habituate the patient's associated negative emotional reactions (annoyance) to tinnitus, its perception (awareness) and, ultimately, its impact on the participant's life. Study participants will include active and retired military personnel of the U. S. Armed Forces and their dependents who suffer from severe tinnitus. The study will be conducted at flagship Air Force, and Navy Medical Centers.

This trial will evaluate the efficacy of TRT and its components (DC and ST) versus the standard of care (SC) as administered in the military by comparing the efficacy of:

* (1) TRT (DC and ST achieved using conventional sound generators) versus SC;
* (2) TRT versus partial TRT (DC and placebo sound generators) to evaluate the separate effect of sound therapy, under the assumption that placebo noise generator will not provide any meaningful sound therapy beyond that found in SC;
* (3) partial TRT versus SC to evaluate the separate effect of DC.

Eligibility will be determined at the Baseline Eligibility Visit, which will consist of a medical and tinnitus history, physical examination, and baseline audiological/tinnitus/hyperacusis evaluation. Study participants will also complete a series of quality of life and psychological profile tests. Study Audiologists will administer the randomly assigned treatment. Follow-up visits at Clinical Centers will take place at 3, 6, 12, and 18 months and include completion of tinnitus outcome questionnaires at all visits. Psychometric testing and audiological/tinnitus/hyperacusis evaluation will take place at the 6, 12, and 18 month visits. Evaluation of audiometric pure tone and loudness discomfort level also will take place at treatment visits.

The primary outcome to be measured in the TRTT will be change in scores on the Tinnitus Questionnaire (TQ) longitudinally assessed between baseline and follow-up (i.e., at 3, 6, 12 and 18 months following treatment). Secondary outcomes include changes in the sub-scales of the TQ, change in scores from the Tinnitus Handicap Inventory (THI), Tinnitus Functional Index (TFI), Hearing Handicap Inventory (HHI), and TRT visual analogue scales, and change in the Digit Symbol Substitution Test (DSST). Psychometric secondary outcomes also include change in psychoacoustic variables related to the tinnitus sensation, including tinnitus pitch and loudness match, and loudness discomfort level.

The TRTT is designed to have sufficient power to detect a minimal clinically important difference in the Tinnitus Questionnaire (TQ) i.e., a 10 point difference between TRT and SC groups on change in TQ global scores longitudinally assessed over the course of follow-up and a 7-point difference on TQ score by TRT components, DC and ST.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Subjective severe tinnitus, defined as a score on the Tinnitus Questionnaire (TQ) greater than or equal to 40
* Eligible for care at a Department of Defense Clinical Center
* Speaks English well enough to complete a series of questionnaires and benefit from counseling

Exclusion Criteria:

* Involvement in pending tinnitus-related financial claims or litigation except that associated with usual Veterans' Administration retirement claims
* Tinnitus of less than 12 months duration
* Treatment for tinnitus within previous 12 months
* Routine unavoidable exposure to hazardous noise
* Use of a cancer chemotherapeutic drug within previous 12 months
* Treatment for head or neck injury within previous 24 months
* Treatment for an emotional, psychological, or psychiatric condition within previous 12 months resulting in inability to participate in the trial or complete all followup visits, as assessed by best clinical judgment
* Requirement for use of an ototoxic drug
* Hearing impairment, defined by audiometric thresholds > 30 dB HL at and below 2,000 Hz and > 40 dB HL at 4,000 and 8,000 Hz
* Required use of hearing aids
* Fluctuating hearing loss at a level that would interfere with the reliability of study results
* One or more prominent spontaneous otoacoustic emissions, defined as the presence of a spontaneous otoacoustic emission spike that is 3 or more times larger than the measured variation in amplitude across the remaining frequency range and/or if the emission corresponds in pitch to the tinnitus pitch
* Pulsatile somatosounds suggesting presence of abnormal vasculature or high blood pressure contributing to the tinnitus
* Feigning tinnitus or hearing loss
* Evidence by audiological testing of a treatable etiology of the tinnitus, such as conductive hearing impairment as shown by pure-tone thresholds, abnormal acoustic immittance, abnormal stapedial reflex test, or abnormal auditory brainstem response
* Predisposing disease with tinnitus symptoms amenable to medical or surgical intervention, including but not limited to; chronic otitis media, otosclerosis, vestibular disorder or dizziness, Eustachian tube, middle ear, or inner ear disease, Lyme disease or ear autoimmune disease, malocclusion or temporomandibular joint disease, uncontrolled allergies, aberrant ear, head, or neck blood vasculature or glomus tumor, neurological condition such as multiple sclerosis or ear-related demyelinating disease, perilymphatic fistula, or facial weakness or paralysis
* Meniere's disease
* Uncontrolled diabetes, defined as blood glucose consistently ≥ 200 mg/dl or an HBA1c above 8%
* Evidence from any laboratory study that suggests an etiology for the tinnitus that is treatable, including, but not limited to, abnormal thyroid stimulating hormone (TSH) or thyroid hormone (T3 or T4) levels, positive fluorescent treponemal antibody (FTA) test, or positive Lyme titer
* Evidence of a tumor contributing to the tinnitus, including an acoustic neuroma (or vestibular schwannoma), cerebellopontine angle tumor, skull base tumor, or any other type of tumor that the examining physician believes is responsible for the tinnitus
* Diagnosis of traumatic head or brain injury requiring treatment
* Diagnosis of an emotional, psychological, or psychiatric condition requiring treatment and resulting in inability to participate in the trial or complete all followup visits, as assessed by best clinical judgment
* Inability or unwillingness of patient to comply with study requirements
* Unwillingness of Clinical Center Director to randomize the patient to treatment due to the presence of any condition, physical, mental or social, which is likely to affect the patient returning for follow-up visits on schedule or which is likely to impair his or her performance on the functional tests
* Inability or unwillingness of patient to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Craig Formby, PhD, Study Chair — The University of Alabama, Tuscaloosa; Roberta W Scherer, PhD, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (6):
- United States (6):
  - Naval Hospital Camp Pendleton, Camp Pendleton, California
  - Naval Medical Center, San Diego, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Portsmouth Naval Medical Center, Portsmouth, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Requests for limited datasets may be made to the TRTT Data Coordinating Center

REFERENCES:
- [Background] Scherer RW, Formby C, Gold S, Erdman S, Rodhe C, Carlson M, Shade D, Tucker M, Sensinger LM, Hughes G, Conley GS, Downey N, Eades C, Jylkka M, Haber-Perez A, Harper C, Russell SK, Sierra-Irizarry B, Sullivan M; Tinnitus Retraining Therapy Trial Research Group. The Tinnitus Retraining Therapy Trial (TRTT): study protocol for a randomized controlled trial. Trials. 2014 Oct 15;15:396. doi: 10.1186/1745-6215-15-396. PMID 25319676
- [Background] Formby C, Scherer R; TRTT Study Group. Rationale for the tinnitus retraining therapy trial. Noise Health. 2013 Mar-Apr;15(63):134-42. doi: 10.4103/1463-1741.110299. PMID 23571304
- [Derived] Formby C, Yang X, Scherer RW. Contributions of Counseling and Sound Generator Use in Tinnitus Retraining Therapy: Treatment Response Dynamics Assessed in a Secondary Analysis of a Randomized Trial. J Speech Lang Hear Res. 2022 Feb 9;65(2):816-828. doi: 10.1044/2021_JSLHR-21-00210. Epub 2022 Jan 24. PMID 35073492
- [Derived] Scherer RW, Erdman SA, Gold S, Formby C; TRTT Research Group. Treatment fidelity in the Tinnitus Retraining Therapy Trial. Trials. 2020 Jul 23;21(1):670. doi: 10.1186/s13063-020-04530-9. PMID 32703244
- [Derived] Tinnitus Retraining Therapy Trial Research Group; Scherer RW, Formby C. Effect of Tinnitus Retraining Therapy vs Standard of Care on Tinnitus-Related Quality of Life: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2019 Jul 1;145(7):597-608. doi: 10.1001/jamaoto.2019.0821. PMID 31120533
- [Derived] Scherer RW, Sensinger LD, Sierra-Irizarry B, Formby C; TRTT Research Group. Lessons learned conducting a multi-center trial with a military population: The Tinnitus Retraining Therapy Trial. Clin Trials. 2018 Oct;15(5):429-435. doi: 10.1177/1740774518777709. Epub 2018 May 23. PMID 29792074

RESULTS

PARTICIPANT FLOW:
Groups:
- Tinnitus Retraining Therapy (TRT): TRT includes sound therapy using a conventional sound generator and educational directive counseling (DC).
  The conventional sound generator (SG) is a Tranquil model (General Hearing Instruments, Inc.), worn either inside- or outside-the-ear. The device generates low-level noise and is set at or just below the participant's mixing point (i.e., noise level that just blends with the tinnitus)
  Directive Counseling (DC) involves a one to two-hour educational session during which the participant is given information regarding the nature of the tinnitus problem and related problems such as hearing loss and sound intolerance; visual aids to review the audiological/tinnitus/ hyperacusis evaluation, instruction on anatomy and physiology of hearing and tinnitus, introduction to the Jastreboff neurophysiological model of tinnitus and related concepts of habituation, and use of sound therapy and environmental sound in the habituation process.
- Partial Tinnitus Retraining Therapy (Partial TRT): Partial TRT includes treatment with a placebo sound generator (placebo SG) and directive counseling (DC).
  The placebo sound generator (SG) is a Tranquil model (General Hearing Instruments, Inc.), worn either inside- or outside-the-ear. The device is set at or just below the participant's mixing point (i.e., noise level that just blends with the tinnitus) and generates a low-level sound different from the active devices.
  Directive Counseling (DC) involves a one to two-hour educational session during which the participant is given information regarding the nature of the tinnitus problem and related problems such as hearing loss and sound intolerance; visual aids to review the audiological/tinnitus/ hyperacusis evaluation, instruction on anatomy and physiology of hearing and tinnitus, introduction to the Jastreboff neurophysiological model of tinnitus and related concepts of habituation, and use of sound therapy and environmental sound in the habituation process.
Period: Overall Study
Arm/Group | Tinnitus Retraining Therapy (TRT) | Partial Tinnitus Retraining Therapy (Partial TRT) | Standard of Care (SC)
Started | 51 | 51 | 49
Completed | 41 | 41 | 47
Not Completed | 10 | 10 | 2
Not completed — Withdrawal by Subject | 10 | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tinnitus Retraining Therapy (TRT) | Partial Tinnitus Retraining Therapy (Partial TRT) | Standard of Care (SC) | Total
Number analyzed (Participants) | 51 | 51 | 49 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (12.6) | 50.9 (11.2) | 49.9 (10.6) | 50.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 13 | 44
  Male | 34 | 37 | 36 | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 5 | 6 | 7 | 18
  White | 36 | 39 | 35 | 110
  More than one race | 4 | 0 | 3 | 7
  Unknown or Not Reported | 2 | 1 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 5 | 17
  Not Hispanic or Latino | 41 | 44 | 41 | 126
  Unknown or not reported | 3 | 2 | 3 | 8
Marital status [Count of Participants; unit: Participants]
  Married/living with partner | 39 | 41 | 41 | 121
  Single/never married | 4 | 6 | 3 | 13
  Divorced/separated | 7 | 4 | 4 | 15
  Widowed | 0 | 0 | 1 | 1
  Other/unknown | 1 | 0 | 0 | 1
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 0 | 3 | 2 | 5
  Previous smoker | 15 | 15 | 11 | 41
  Never smoked | 36 | 33 | 36 | 105
Duration of tinnitus as a problem [Count of Participants; unit: Participants]
  Less than 2 years | 12 | 11 | 6 | 29
  More than 2 years but less than 5 years | 15 | 17 | 20 | 52
  More than 5 years | 24 | 22 | 22 | 68
  Unknown/missing | 0 | 1 | 1 | 2
Tinnitus type of sound [Count of Participants; unit: Participants]
  Tonal (ringing, music, whistling, etc.) | 47 | 47 | 47 | 141
  Low frequency (buzzing, puldating, ocean, etc. | 4 | 2 | 1 | 7
  High frequency (hissing, sizzling, ectc.) | 0 | 1 | 0 | 1
  Other (clicking, crickets, etc.) | 0 | 1 | 0 | 1
  Missing | 0 | 0 | 1 | 1
Tinnitus location [Count of Participants; unit: Participants]
  One ear | 11 | 4 | 4 | 19
  Both ears | 22 | 24 | 20 | 66
  In the head | 7 | 11 | 10 | 28
  In the head and one or both ears | 11 | 12 | 15 | 38
Baseline scores on the Tinnitus Questionnaire and sub-scales [Mean (Standard Deviation); unit: units on a scale] — The Tinnitus Questionnaire has 52 questions, scored as 0, 1, or 2. The total score is the sum of the scores of all questions and ranges from 0 to 102, with higher scores indicating more tinnitus distress. Sub-scales (range of scores) include auditory perceptual difficulties (0 to 14), emotional distress (0 to 38), intrusiveness (0 to 14), sleep disturbance (0 to 8), and somatic complaint (0 to 8).
  units on a scale
    Total | 56.4 (11.9) | 54.4 (11.5) | 54.6 (11.2) | 55.1 (11.5)
    Auditory perceptual | 7.2 (2.8) | 7.1 (3.0) | 7.7 (3.7) | 7.3 (3.1)
    Emotional distress | 17.2 (6.2) | 17.0 (6.6) | 15.8 (5.5) | 16.7 (6.1)
    Intrusiveness | 9.9 (2.0) | 9.9 (2.1) | 9.8 (1.8) | 9.9 (2.0)
    Sleep disturbance | 4.9 (2.3) | 4.3 (2.2) | 4.8 (2.4) | 4.7 (2.3)
    Somatic complaint | 5.3 (1.6) | 4.5 (1.8) | 4.9 (1.7) | 4.9 (1.7)
Baseline scores on Tinnitus Functional Index and sub-scales [Mean (Standard Deviation); unit: units on a scale] — The Tinnitus Functional Index (TFI) has 25 questions, scored from 0 to 10. The total score ranges from 0 to 100, with higher scores indicating more tinnitus distress. All sub-scales are normalized to range from 0 to 100 scores. Sub-scales include auditory difficulties, cognitive interference, emotional distress, intrusiveness, reduced sense of control, reduced quality of life, relaxation interference, and sleep disturbance.
  units on a scale
    Total | 48.1 (17.6) | 50.3 (17.1) | 53.5 (17.3) | 50.6 (17.3)
    Auditory difficulties | 45.1 (27.2) | 45.0 (27.2) | 46.6 (25.7) | 45.6 (25.9)
    Cognitive interference | 42.7 (21.2) | 51.0 (22.1) | 47.8 (24.5) | 47.2 (22.7)
    Emotional distress | 31.6 (24.6) | 31.8 (26.1) | 34.4 (23.6) | 32.6 (24.7)
    Intrusiveness | 63.3 (23.2) | 67.5 (18.0) | 70.7 (17.3) | 67.1 (19.8)
    Reduced sense of control | 58.6 (20.9) | 63.7 (16.7) | 67.8 (19.5) | 63.3 (19.3)
    Reduced quality of life | 30.1 (22.7) | 35.7 (23.1) | 37.0 (25.4) | 34.2 (23.8)
    Relaxation difficulties | 63.9 (23.6) | 61.9 (27.2) | 68.2 (24.4) | 64.6 (25.1)
    Sleep disturbance | 55.4 (30.8) | 50.3 (28.1) | 61.0 (30.2) | 55.5 (29.8)
Baseline scores on the Tinnitus Handicap Inventory and sub-scales [Mean (Standard Deviation); unit: units on a scale] — The Tinnitus Handicap Inventory has 25 questions scored as 0, 2, or 4 for "no", "sometimes", and "yes" respectively for a total score ranging from 0 to 100, with higher scores indicated more tinnitus distress. Subscales (ranges for scores) are functional (0 to 44), emotional (0 to 36) and catastrophic (0 to 20).
  units on a scale
    Total | 37.8 (13.0) | 42.3 (20.7) | 38.6 (16.7) | 39.6 (17.1)
    Functional subscale | 18.4 (6.2) | 20.9 (9.5) | 19.3 (8.4) | 19.5 (8.2)
    Emotional subscale | 11.3 (6.2) | 12.7 (9.0) | 11.4 (7.1) | 11.8 (7.5)
    Catastrophic subscale | 8.2 (3.4) | 8.7 (4.2) | 8.0 (3.5) | 8.3 (3.7)
Rank of tinnitus as problem [Mean (Standard Deviation); unit: units on a scale] — The question "How much of a problem is tinnitus?" was scored on a visual analogue scale from 0 ("no problem at all") to 10 "as much as you can imagine".
  units on a scale | 6.2 (2.2) | 6.4 (2.2) | 6.3 (2.1) | 6.3 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Tinnitus Questionnaire (TQ) From Baseline to 3, 6, 12, and 18 Months
Description: The TQ is a tinnitus-specific health-related quality of life instrument with 52 statements that the respondent marks as true, partly true, or not true. The TQ is scored from 0 to 102, with higher scores indicating more of an impact of the tinnitus on quality of life. Subscales include emotional distress, intrusiveness, auditory perceptual difficulties, sleep disturbance,and somatic complaints.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy (TRT) | Partial Tinnitus Retraining Therapy (Partial TRT) | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 37 | 42
  Change from baseline to 3 months | -17.8 (13.6) | -15.4 (15.9) | -11.5 (13.4)
  Change from baseline to 6 months: number analyzed (Participants) | 32 | 35 | 38
  Change from baseline to 6 months | -22.0 (15.6) | -18.3 (15.4) | -14.5 (14.8)
  Change from baseline to 12 months: number analyzed (Participants) | 34 | 30 | 30
  Change from baseline to 12 months | -21.1 (15.1) | -21.8 (15.9) | -17.6 (14.0)
  Change from baseline to 18 months: number analyzed (Participants) | 34 | 40 | 37
  Change from baseline to 18 months | -18.2 (15.2) | -19.0 (15.9) | -16.5 (16.3)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy (TRT) vs Standard of Care (SC); Test type: Superiority; p = 0.47, repeated measures GEE model — The a priori threshold for statistical significance was <0.025 to account for two comparisons: (1) TRT versus the Standard of Care and (2) Partial TRT versus the Standard of Care; Slope = -2.35, 95% CI 2-sided [-8.77 to 4.07], Standard Error of Mean 3.27 — Adjusted for baseline TQ value, clinic, visit, age, gender, baseline Positive and Negative Affect Schedule and State Trait Anxiety Inventory scores, with multiple imputation
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy (Partial TRT) vs Standard of Care (SC); Test type: Superiority; p = 0.31, repeated measures GEE model — [p-value comment as in outcome 1, analysis 1]; Slope = -2.80, 95% CI 2-sided [-8.27 to 2.65], Standard Error of Mean 2.78 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change in Tinnitus Functional Index (TFI) From Baseline to 3, 6, 12, and 18 Months
Description: The TFI is a tinnitus-specific health -related quality of life instrument. Subscales include intrusiveness, reduced sense of control, cognitive interference, sleep disturbance, auditory difficulties (related to tinnitus), relaxation interference, reduced quality of life, and emotional distress. The total and each subscale score ranges from 0 to 100 with higher scores indicated a greater impact of tinnitus on quality of life.
Time Frame: Baseline and 3, 6, 12, and 18 months
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy (TRT) | Partial Tinnitus Retraining Therapy (Partial TRT) | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | -3.7 (15.3) | -10.9 (18.0) | -4.4 (12.7)
  Change from baseline to 6 months: number analyzed (Participants) | 32 | 35 | 38
  Change from baseline to 6 months | -9.6 (14.2) | -9.5 (18.6) | -8.7 (18.0)
  Change from baseline to 12 months: number analyzed (Participants) | 34 | 30 | 30
  Change from baseline to 12 months | -7.7 (18.6) | -17.2 (17.7) | -16.3 (19.2)
  Change from baseline to 18 months: number analyzed (Participants) | 34 | 40 | 37
  Change from baseline to 18 months | -6.7 (18.5) | -14.4 (17.2) | -10.3 (21.9)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy (TRT) vs Standard of Care (SC); Test type: Superiority; p = 0.96, repeated measures GEE model — The a priori threshold for statistical significance was <0.025 to account for two comparisons: (1) TRT versus the Standard of Care and (2) Partial TRT versus the Standard of Ca; Slope = -0.14, 95% CI 2-sided [-5.30 to 5.02], Standard Error of Mean 2.63 — Adjusted for baseline TFI value, clinic, visit, age, gender, baseline Positive and Negative Affect Schedule and State Trait Anxiety Inventory scores, with multiple imputation
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy (Partial TRT) vs Standard of Care (SC); Test type: Superiority; p = 0.28, repeated measures GEE model — The a priori threshold for statistical significance was <0.025 to adjust for two comparisons: (1) TRT versus the Standard of Care and (2) Partial TRT versus the Standard of Ca; Slope = 2.74, 95% CI 2-sided [-2.21 to 7.70], Standard Error of Mean 2.53 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Change in Tinnitus Handicap Inventory (THI) Score From Baseline to 3, 6, 12, and 18 Months Follow-up
Description: Change in THI score from baseline to 3 months follow-up. The THI is a tinnitus-specific health-related quality of life instrument. Subscales include the functional (scored 0 to 44), emotional (scored 0 to 36) and catastrophic (scored 0 to 20). The total score ranges from 0 to 100 with higher scores indicating a greater impact of tinnitus on quality of life.
Time Frame: Baseline and 3. 6. 12. and 18 months
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy (TRT) | Partial Tinnitus Retraining Therapy (Partial TRT) | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | -6.0 (15.8) | -13.6 (18.4) | -2.9 (13.6)
  Change from baseline to 6 months: number analyzed (Participants) | 31 | 35 | 38
  Change from baseline to 6 months | -10.3 (12.8) | -11.0 (19.1) | -5.3 (20.6)
  Change from baseline to 12 months: number analyzed (Participants) | 33 | 28 | 30
  Change from baseline to 12 months | -7.4 (16.3) | -14.9 (17.2) | -12.0 (15.5)
  Change from baseline to 18 months: number analyzed (Participants) | 33 | 39 | 37
  Change from baseline to 18 months | -6.1 (18.0) | -12.6 (17.1) | -9.4 (17.7)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy (TRT) vs Standard of Care (SC); Test type: Superiority; p = 0.30, repeated measures GEE model — [p-value comment as in outcome 1, analysis 1]; Slope = 0.61, 95% CI 2-sided [-0.55 to 1.77], Standard Error of Mean 0.59 — Adjusted for baseline THI value, clinic, visit, age, gender, baseline Positive and Negative Affect Schedule and State Trait Anxiety Inventory scores, with multiple imputation
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy (Partial TRT) vs Standard of Care (SC); Test type: Superiority; p = 0.29, repeated measures GEE model — [p-value comment as in outcome 2, analysis 1]; Slope = -0.62, 95% CI 2-sided [-1.75 to 0.52], Standard Error of Mean 0.58 — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change in Tinnitus Retraining Therapy Interview Visual Analogue Scales at 3, 6, 12, and 18 Months Follow-up
Description: 10 point visual analog scale asking "How much of a problem is tinnitus?" on a scale from 0 "no problem at all" to 10 "as much as you can imagine"
Time Frame: Baseline to 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy (TRT) | Partial Tinnitus Retraining Therapy (Partial TRT) | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 6 months: number analyzed (Participants) | 31 | 35 | 39
  Change from baseline to 6 months | -1.6 (2.4) | -1.4 (2.3) | -1.3 (2.6)
  Change from baseline to 12 months: number analyzed (Participants) | 32 | 26 | 29
  Change from baseline to 12 months | -1.9 (2.6) | -2.0 (2.6) | -2.1 (2.7)
  Change from baseline to 18 months: number analyzed (Participants) | 29 | 30 | 33
  Change from baseline to 18 months | -1.8 (3.0) | -2.1 (2.4) | -1.8 (2.8)

5. Secondary Outcome: Change in Tinnitus Questionnaire Emotional Distress Sub-scale Scores From Baseline to 3, 6, 12, and 18 Months.
Description: Change in Tinnitus Questionnaire emotional distress sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 38 with higher scores representing greater emotional distress.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tinnitus Retraining Therapy: TRT includes sound therapy using a conventional sound generator and educational directive counseling (DC).
  The conventional sound generator (SG) is a Tranquil model (General Hearing Instruments, Inc.), worn either inside- or outside-the-ear. The device generates low-level noise and is set at or just below the participant's mixing point (i.e., noise level that just blends with the tinnitus)
  Directive Counseling (DC) involves a one to two-hour educational session during which the participant is given information regarding the nature of the tinnitus problem and related problems such as hearing loss and sound intolerance; visual aids to review the audiological/tinnitus/ hyperacusis evaluation, instruction on anatomy and physiology of hearing and tinnitus, introduction to the Jastreboff neurophysiological model of tinnitus and related concepts of habituation, and use of sound therapy and environmental sound in the habituation process.
- Partial Tinnitus Retraining Therapy: Partial TRT includes treatment with a placebo sound generator (placebo SG) and directive counseling (DC).
  Placebo sound generator (placebo SG): Tranquil model placebo sound generators (General Hearing Instruments, Inc.) are either inside or outside-the-ear devices that generate a sound different from the active devices.
  Directive Counseling (DC): two-hour educational session during which the patient is given information regarding the nature of the tinnitus problem and related problems such as hearing loss and sound intolerance; visual aids to review the audiological/tinnitus/ hyperacusis evaluation, provide instruction on anatomy and physiology of hearing and tinnitus, introduce the Jastreboff neurophysiological model of tinnitus and related concepts of habituation, and describe and recommend the use of ST and environmental sound in the habituation process.
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 37 | 42
  Change from baseline to 3 months | -7.2 (6.3) | -6.6 (8.0) | -4.6 (6.2)
  Change from baseline to 6 months: number analyzed (Participants) | 31 | 35 | 38
  Change from baseline to 6 months | -8.8 (6.8) | -7.8 (8.3) | -6.0 (6.5)
  Change from baseline to 12 months: number analyzed (Participants) | 33 | 29 | 30
  Change from baseline to 12 months | -8.9 (6.4) | -9.0 (7.0) | -7.4 (5.8)
  Change from baseline to 18 months: number analyzed (Participants) | 33 | 39 | 37
  Change from baseline to 18 months | -8.1 (6.3) | -8.7 (7.9) | -7.4 (6.3)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.77, repeated measures GEE model — The a priori threshold for statistical significance was <0.025 to account for two comparisons (1) TRT versus the Standard of Care and (2) Partial TRT versus the Standard of Care; Slope = -0.39, 95% CI 2-sided [-3.08 to 2.29], Standard Error of Mean 1.37 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.65, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -0.60, 95% CI 2-sided [-3.16 to 1.96], Standard Error of Mean 1.30 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change in Tinnitus Questionnaire Intrusiveness Sub-scale Scores.
Description: Change in Tinnitus Questionnaire intrusiveness sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 14 with higher scores representing greater intrusiveness of the tinnitus.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 37 | 42
  Change from baseline to 3 months | -2.4 (3.3) | -1.7 (2.8) | -1.4 (2.5)
  Change from baseline to 6 months: number analyzed (Participants) | 31 | 35 | 38
  Change from baseline to 6 months | -2.2 (2.7) | -2.2 (3.1) | -2.0 (3.2)
  Change from baseline to 12 months: number analyzed (Participants) | 33 | 29 | 30
  Change from baseline to 12 months | -3.0 (3.0) | -3.1 (3.0) | -2.2 (3.3)
  Change from baseline to 18 months: number analyzed (Participants) | 33 | 39 | 37
  Change from baseline to 18 months | -3.2 (3.3) | -2.4 (2.9) | -2.4 (3.3)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.50, repeated measures GEE model — The a priori threshold for statistical significance was set at <0.025 to account for two comparisons (1) TRT versus the Standard of Care and (2) Partial TRT versus the Standard of Care; Slope = -0.36, 95% CI 2-sided [-1.38 to 0.67], Standard Error of Mean 0.52 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.82, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -0.12, 95% CI 2-sided [-1.14 to 0.90], Standard Error of Mean 0.52 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change in Tinnitus Questionnaire Auditory Perceptual Difficulties Sub-scale Scores.
Description: Change in Tinnitus Questionnaire auditory perceptual sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 14 with higher scores representing greater auditory difficulties.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including all data from participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 37 | 42
  Change from baseline to 3 months | -2.5 (2.6) | -1.8 (3.0) | -1.2 (2.5)
  Change from baseline to 6 months: number analyzed (Participants) | 31 | 35 | 38
  Change from baseline to 6 months | -2.4 (2.9) | -2.4 (2.6) | -2.1 (3.2)
  Change from baseline to 12 months: number analyzed (Participants) | 33 | 29 | 30
  Change from baseline to 12 months | -2.6 (2.4) | -2.3 (2.9) | -2.6 (3.0)
  Change from baseline to 18 months: number analyzed (Participants) | 33 | 39 | 37
  Change from baseline to 18 months | -2.0 (3.0) | -2.0 (3.2) | -2.4 (3.2)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.46, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -0.38, 95% CI 2-sided [-1.37 to 0.62], Standard Error of Mean 0.51 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority — The a priori threshold for statistical significance was <0.025 to account for two comparisons (1) TRT versus the Standard of Care and (2) Partial TRT versus the Standard of Care; p = 0.48, repeated measures GEE model; Slope = -0.36, 95% CI 2-sided [-1.35 to 0.64], Standard Error of Mean 0.51 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change in Tinnitus Questionnaire Sleep Disturbance Sub-scale Scores.
Description: Change in Tinnitus Questionnaire sleep disturbance sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 8 with higher scores representing greater sleep disturbance.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 37 | 42
  Change from baseline to 3 months | -1.4 (1.7) | -1.9 (2.2) | -1.2 (1.7)
  Change from baseline to 6 months: number analyzed (Participants) | 31 | 35 | 38
  Change from baseline to 6 months | -1.7 (2.0) | -1.8 (1.9) | -1.2 (1.7)
  Change from baseline to 12 months: number analyzed (Participants) | 33 | 29 | 30
  Change from baseline to 12 months | -1.7 (2.4) | -2.3 (2.5) | -1.4 (1.9)
  Change from baseline to 18 months: number analyzed (Participants) | 33 | 39 | 37
  Change from baseline to 18 months | -1.6 (2.3) | -2.2 (2.0) | -1.2 (2.1)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.75, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -0.10, 95% CI 2-sided [-0.74 to 0.53], Standard Error of Mean 0.32 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.015, repeated measures GEE model — The a priori threshold for statistical significance was < 0.025 to account for two comparisons (1) TRT versus the Standard of Care and (2) Partial TRT versus the Standard of Care; Slope = -0.87, 95% CI 2-sided [-1.56 to -0.17], Standard Error of Mean 0.35 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change in Tinnitus Questionnaire Somatic Complaint Sub-scale Scores.
Description: Change in Tinnitus Questionnaire somatic complaint sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 8 with higher scores representing greater somatic complaints.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 37 | 42
  Change from baseline to 3 months | -1.9 (2.0) | -1.2 (1.9) | -1.2 (2.1)
  Change from baseline to 6 months: number analyzed (Participants) | 31 | 35 | 38
  Change from baseline to 6 months | -2.2 (1.7) | -1.6 (1.8) | -1.5 (2.0)
  Change from baseline to 12 months: number analyzed (Participants) | 33 | 29 | 33
  Change from baseline to 12 months | -2.1 (1.8) | -1.7 (2.0) | -1.6 (2.0)
  Change from baseline to 18 months: number analyzed (Participants) | 33 | 39 | 37
  Change from baseline to 18 months | -1.7 (1.9) | -1.5 (2.1) | -1.3 (2.1)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.85, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -0.07, 95% CI 2-sided [-0.83 to 0.69], Standard Error of Mean 0.39 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.55, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -0.20, 95% CI 2-sided [-0.86 to 0.46], Standard Error of Mean 0.34 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change in Tinnitus Functional Index Intrusiveness Sub-scale Scores.
Description: Change in Tinnitus Functional Index intrusiveness sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 100 with higher scores representing greater intrusiveness of the tinnitus.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | -1.9 (21.7) | -6.3 (19.7) | -2.9 (17.9)
  Change from baseline to 6 months: number analyzed (Participants) | 32 | 35 | 38
  Change from baseline to 6 months | -11.9 (17.9) | -8.8 (22.2) | -10.4 (21.7)
  Change from baseline to 12 months: number analyzed (Participants) | 34 | 30 | 30
  Change from baseline to 12 months | -8.1 (26.2) | -16.6 (21.3) | -19.4 (25.2)
  Change from baseline to 18 months: number analyzed (Participants) | 34 | 40 | 37
  Change from baseline to 18 months | -6.8 (27.8) | -10.1 (20.6) | -11.4 (26.4)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.30, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -3.19, 95% CI 2-sided [-9.27 to 2.88], Standard Error of Mean 3.10 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.76, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -0.91, 95% CI 2-sided [-6.75 to 4.93], Standard Error of Mean 2.98 — [estimate comment as in outcome 2, analysis 1]

11. Secondary Outcome: Change in Tinnitus Functional Index Reduced Sense of Control Sub-scale Scores.
Description: Change in Tinnitus Functional Index reduced sense of control sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 100 with higher scores representing greater reduction of control.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | 0.2 (19.0) | -9.2 (23.6) | -9.4 (17.0)
  Change from baseline to 6 months: number analyzed (Participants) | 32 | 35 | 38
  Change from baseline to 6 months | -8.0 (18.5) | -7.0 (24.9) | -12.4 (22.1)
  Change from baseline to 12 months: number analyzed (Participants) | 34 | 30 | 30
  Change from baseline to 12 months | -6.6 (20.1) | -20.8 (25.1) | -25.3 (24.7)
  Change from baseline to 18 months: number analyzed (Participants) | 34 | 40 | 37
  Change from baseline to 18 months | -9.0 (21.5) | -12.0 (24.0) | -20.5 (27.6)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.35, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = 3.12, 95% CI 2-sided [-3.44 to 9.68], Standard Error of Mean 3.34 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.30, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = 3.29, 95% CI 2-sided [-2.96 to 9.54], Standard Error of Mean 3.19 — [estimate comment as in outcome 2, analysis 1]

12. Secondary Outcome: Change in Tinnitus Functional Index Cognitive Interference Sub-scale Scores.
Description: Change in Tinnitus Functional Index cognitive interference sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 100 with higher scores representing greater cognitive interference.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | -2.2 (20.0) | -13.1 (22.5) | -3.0 (21.2)
  Change from baseline to 6 months: number analyzed (Participants) | 32 | 35 | 38
  Change from baseline to 6 months | -7.5 (17.3) | -12.2 (23.3) | -6.7 (22.4)
  Change from baseline to 12 months: number analyzed (Participants) | 34 | 30 | 30
  Change from baseline to 12 months | -2.4 (21.4) | -15.4 (21.4) | -9.1 (24.5)
  Change from baseline to 18 months: number analyzed (Participants) | 34 | 40 | 37
  Change from baseline to 18 months | -1.1 (22.2) | -14.7 (21.2) | -8.3 (29.2)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.68, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = 1.41, 95% CI 2-sided [-5.20 to 8.02], Standard Error of Mean 3.37 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.77, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = 0.94, 95% CI 2-sided [-5.44 to 7.33], Standard Error of Mean 3.26 — [estimate comment as in outcome 2, analysis 1]

13. Secondary Outcome: Change in Tinnitus Functional Index Sleep Disturbance Sub-scale Scores.
Description: Change in Tinnitus Functional Index sleep disturbance sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 100 with higher scores representing greater sleep disturbance.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | -7.2 (23.9) | -16.1 (24.9) | -4.0 (21.1)
  Change from baseline to 6 months: number analyzed (Participants) | 32 | 35 | 38
  Change from baseline to 6 months | -13.0 (27.3) | -10.8 (28.4) | -11.2 (23.5)
  Change from baseline to 12 months: number analyzed (Participants) | 34 | 30 | 30
  Change from baseline to 12 months | -10.9 (27.7) | -20.6 (26.9) | -15.9 (29.0)
  Change from baseline to 18 months: number analyzed (Participants) | 34 | 40 | 37
  Change from baseline to 18 months | -11.1 (31.4) | -20.2 (23.4) | -10.0 (24.3)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.43, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -3.53, 95% CI 2-sided [-12.30 to 5.23], Standard Error of Mean 4.47 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.001, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -13.70, 95% CI 2-sided [-22.02 to -5.38], Standard Error of Mean 4.24 — [estimate comment as in outcome 2, analysis 1]

14. Secondary Outcome: Change in Tinnitus Functional Index Auditory Difficulties Sub-scale Scores.
Description: Change in Tinnitus Functional Index auditory difficulties sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 100 with higher scores representing greater auditory difficulties.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | 0.3 (26.0) | -8.9 (24.5) | 1.2 (21.3)
  Change from baseline to 6 months: number analyzed (Participants) | 32 | 35 | 38
  Change from baseline to 6 months | -5.3 (21.8) | -3.8 (28.3) | -2.5 (33.7)
  Change from baseline to 12 months: number analyzed (Participants) | 34 | 30 | 30
  Change from baseline to 12 months | -7.9 (24.3) | -13.2 (24.9) | -11.8 (29.2)
  Change from baseline to 18 months: number analyzed (Participants) | 34 | 40 | 37
  Change from baseline to 18 months | -7.1 (21.1) | -6.6 (22.3) | -2.7 (29.2)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.34, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = 3.71, 95% CI 2-sided [-3.96 to 11.38], Standard Error of Mean 3.91 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.95, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -0.23, 95% CI 2-sided [-7.72 to 7.26], Standard Error of Mean 3.82 — [estimate comment as in outcome 2, analysis 1]

15. Secondary Outcome: Change in Tinnitus Functional Index Relaxation Interference Sub-scale Scores.
Description: Change in Tinnitus Functional Index relaxation interference sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 100 with higher scores representing greater relaxation interference.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | -7.6 (24.3) | -12.9 (26.7) | -4.6 (24.8)
  Change from baseline to 6 months: number analyzed (Participants) | 32 | 35 | 38
  Change from baseline to 6 months | -12.8 (18.5) | -12.8 (27.8) | -9.6 (24.9)
  Change from baseline to 12 months: number analyzed (Participants) | 34 | 30 | 30
  Change from baseline to 12 months | -16.1 (23.5) | -16.3 (28.1) | -20.3 (33.5)
  Change from baseline to 18 months: number analyzed (Participants) | 34 | 40 | 37
  Change from baseline to 18 months | -13.3 (26.7) | -18.6 (30.2) | -15.6 (33.1)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.62, repeated measures GEE model — [p-value comment as in outcome 8, analysis 2]; Slope = -1.85, 95% CI 2-sided [-9.07 to 5.38], Standard Error of Mean 3.69 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.21, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -4.46, 95% CI 2-sided [-11.48 to 2.55], Standard Error of Mean 3.58 — [estimate comment as in outcome 2, analysis 1]

16. Secondary Outcome: Change in Tinnitus Functional Index Emotional Distress Sub-scale Scores.
Description: Change in Tinnitus Functional Index emotional distress sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 100 with higher scores representing greater emotional distress.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | -6.5 (18.7) | -11.4 (22.1) | -8.1 (16.7)
  Change from baseline to 6 months: number analyzed (Participants) | 32 | 35 | 38
  Change from baseline to 6 months | -12.4 (25.6) | -9.4 (19.8) | -10.0 (26.1)
  Change from baseline to 12 months: number analyzed (Participants) | 34 | 30 | 30
  Change from baseline to 12 months | -7.1 (25.0) | -18.2 (22.1) | -16.9 (22.7)
  Change from baseline to 18 months: number analyzed (Participants) | 34 | 40 | 37
  Change from baseline to 18 months | -7.5 (25.7) | -15.9 (23.5) | -8.8 (28.6)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.97, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -0.13, 95% CI 2-sided [-6.78 to 6.52], Standard Error of Mean 3.39 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.36, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -3.02, 95% CI 2-sided [-9.43 to 3.40], Standard Error of Mean 3.27 — [estimate comment as in outcome 2, analysis 1]

17. Secondary Outcome: Change in Tinnitus Functional Index Reduced Quality of Life Sub-scale Scores.
Description: Change in Tinnitus Functional Index reduced quality of life sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 100 with higher scores representing greater reduction in quality of life.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | -4.6 (19.3) | -12.0 (21.2) | -4.6 (15.5)
  Change from baseline to 6 months: number analyzed (Participants) | 32 | 35 | 38
  Change from baseline to 6 months | -7.0 (18.0) | -10.7 (20.9) | -7.6 (23.7)
  Change from baseline to 12 months: number analyzed (Participants) | 34 | 30 | 30
  Change from baseline to 12 months | -3.7 (22.9) | -16.8 (21.7) | -12.8 (22.8)
  Change from baseline to 18 months: number analyzed (Participants) | 34 | 40 | 37
  Change from baseline to 18 months | -0.3 (23.0) | -16.6 (20.9) | -6.4 (24.4)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.68, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = 1.24, 95% CI 2-sided [-4.67 to 7.14], Standard Error of Mean 3.01 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.23, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -3.52, 95% CI 2-sided [-9.26 to 2.23], Standard Error of Mean 2.93 — [estimate comment as in outcome 2, analysis 1]

18. Secondary Outcome: Change in Tinnitus Handicap Inventory Functional Sub-scale Scores.
Description: Change in Tinnitus Handicap Inventory functional sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 44 with higher scores representing greater functional difficulties.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | -1.3 (7.9) | -6.2 (8.7) | 0.5 (7.5)
  Change from baseline to 6 months: number analyzed (Participants) | 31 | 35 | 38
  Change from baseline to 6 months | -3.2 (6.4) | -4.1 (9.0) | -1.2 (9.3)
  Change from baseline to 12 months: number analyzed (Participants) | 33 | 28 | 30
  Change from baseline to 12 months | -2.2 (7.2) | -6.6 (7.5) | -4.0 (8.0)
  Change from baseline to 18 months: number analyzed (Participants) | 33 | 39 | 37
  Change from baseline to 18 months | -1.5 (8.7) | -5.1 (7.0) | -2.4 (9.7)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.52, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -0.82, 95% CI 2-sided [-3.30 to 1.66], Standard Error of Mean 1.27 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.022, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -2.81, 95% CI 2-sided [-5.21 to -0.41], Standard Error of Mean 1.22 — [estimate comment as in outcome 3, analysis 1]

19. Secondary Outcome: Change in Tinnitus Handicap Inventory Emotional Sub-scale Scores.
Description: Change in Tinnitus Handicap Inventory emotional sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 36 with higher scores representing greater emotional distress.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | -3.0 (6.7) | -4.2 (6.9) | -1.7 (5.4)
  Change from baseline to 6 months: number analyzed (Participants) | 31 | 35 | 38
  Change from baseline to 6 months | -4.1 (5.9) | -4.2 (7.3) | -2.4 (8.5)
  Change from baseline to 12 months: number analyzed (Participants) | 33 | 28 | 30
  Change from baseline to 12 months | -3.3 (7.1) | -4.9 (6.3) | -5.3 (6.3)
  Change from baseline to 18 months: number analyzed (Participants) | 33 | 39 | 37
  Change from baseline to 18 months | -2.8 (8.0) | -4.4 (7.7) | -4.3 (6.2)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.72, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = 0.34, 95% CI 2-sided [-1.54 to 2.23], Standard Error of Mean 0.96 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.26, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -1.04, 95% CI 2-sided [-2.83 to 0.75], Standard Error of Mean 0.91 — [estimate comment as in outcome 3, analysis 1]

20. Secondary Outcome: Change in Tinnitus Handicap Inventory Catastrophic Sub-scale Scores.
Description: Change in Tinnitus Handicap Inventory catastrophic sub-scale from baseline to follow-up. Sub-scale scores range from 0 to 20 with higher scores representing greater catastrophic effect of the tinnitus.
Time Frame: Baseline to 3, 6, 12, and 18 months follow-up
Population: Intention to treat, including data from all participants with at least one follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tinnitus Retraining Therapy | Partial Tinnitus Retraining Therapy | Standard of Care (SC)
Number analyzed (Participants) | 44 | 46 | 46
units on a scale
  Change from baseline to 3 months: number analyzed (Participants) | 40 | 38 | 42
  Change from baseline to 3 months | -1.7 (3.6) | -3.2 (4.8) | -1.8 (3.4)
  Change from baseline to 6 months: number analyzed (Participants) | 31 | 35 | 38
  Change from baseline to 6 months | -3.0 (3.3) | -2.7 (4.7) | -1.8 (4.9)
  Change from baseline to 12 months: number analyzed (Participants) | 33 | 28 | 30
  Change from baseline to 12 months | -1.9 (4.1) | -3.5 (4.7) | -2.7 (3.2)
  Change from baseline to 18 months: number analyzed (Participants) | 33 | 39 | 37
  Change from baseline to 18 months | -1.7 (3.8) | -3.2 (4.4) | -2.7 (4.3)
Statistical Analysis 1: Comparison: Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.30, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = 0.61, 95% CI 2-sided [0.55 to 1.78], Standard Error of Mean 0.59 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Partial Tinnitus Retraining Therapy vs Standard of Care (SC); Test type: Superiority; p = 0.29, repeated measures GEE model — [p-value comment as in outcome 5, analysis 1]; Slope = -0.62, 95% CI 2-sided [-1.75 to 0.52], Standard Error of Mean 0.58 — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to the end of the 18 month follow-up period.
Description: The only adverse event systematically collected was depression, assessed as a score of 4 or more or endorsement of suicidal ideation on the Beck Depression Inventory Short Form. This instrument was administered at each study visit (baseline, 3, 6, 12, and 18 months follow-up).
  Other adverse events were not systematically collected, but reported at the time of incidence.
Arm/Group | Tinnitus Retraining Therapy (TRT) | Partial Tinnitus Retraining Therapy (Partial TRT) | Standard of Care (SC)
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/51 | 3/51 | 0/49
Other Adverse Events (participants affected / at risk) | 10/51 | 12/51 | 9/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tinnitus Retraining Therapy (TRT) (N=51) | Partial Tinnitus Retraining Therapy (Partial TRT) (N=51) | Standard of Care (SC) (N=49)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) — Unspecified cancer
Surgery (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Surgery due to blood clot compressing cerebellum
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tinnitus Retraining Therapy (TRT) (N=51) | Partial Tinnitus Retraining Therapy (Partial TRT) (N=51) | Standard of Care (SC) (N=49)
Depression (Psychiatric disorders) | 9 (12) | 11 (21) | 9 (9) — Score of 4 of more on Beck Depression Inventory at any visit
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0
Pain and swollen ear canal (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) — No redness or oozing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-06-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT01177137/Prot_SAP_ICF_000.pdf